CLINICAL TRIAL: NCT02655354
Title: A Policy Relevant US Trauma Care System Pragmatic Trial for PTSD and Comorbidity
Acronym: TSOS6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Douglas Zatzick, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20150987; UH3MH106338 (NIH)
Record Dates: First submitted 2015-07-27; First posted 2016-01-14 (Estimated); Results first posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Posttraumatic Stress Disorder; Depression; Alcohol-Related Disorders; Suicidal Ideation; Substance-Related Disorders; Mild Cognitive Impairment; Quality of Life; Pain; Wounds and Injury; Brain Injuries; Chronic Disease
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Alcohol-Related Disorders; Suicidal Ideation; Substance-Related Disorders; Cognitive Dysfunction; Pain; Wounds and Injuries; Brain Injuries; Chronic Disease | interventions — Motivational Interviewing; Fluoxetine; Fluvoxamine; Paroxetine; Sertraline; Citalopram; Venlafaxine Hydrochloride; Duloxetine Hydrochloride; Mirtazapine; Diphenhydramine; Trazodone; Prazosin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention aims to prevent the development of chronic PTSD and depressive symptoms, alcohol use problems, and enduring physical disability in survivors of both traumatic brain injury(TBI) and non-TBI injuries. The intervention utilizes a computerized decision support tool to flexibly target these multiple conditions including and includes care management, motivational interviewing, cognitive behavioral therapy elements, psychotropic drugs, and psychotherapy elements.
  Interventions: Behavioral: Motivational Interviewing; Behavioral: Cognitive Behavioral Therapy Elements; Behavioral: Care Management; Drug: Fluoxetine; Drug: Fluvoxamine; Drug: Paroxetine; Drug: Sertraline; Drug: Citalopram; Drug: Venlafaxine; Drug: Duloxetine; Drug: Mirtazapine; Drug: Diphenhydramine; Drug: Trazodone; Drug: Prazosin
- Usual Care (No Intervention): Enhanced standard care practices will be administered to this arm. This enhancement is sharing distressing emotional symptoms at recruitment with the attending nursing staff to address with patient subject.

INTERVENTIONS:
Behavioral: Motivational Interviewing
  Arms: Intervention
Behavioral: Cognitive Behavioral Therapy Elements
  Arms: Intervention
Behavioral: Care Management
  Arms: Intervention
Drug: Fluoxetine — Anti-depressant
  Arms: Intervention
Drug: Fluvoxamine — Anti-depressant
  Arms: Intervention
Drug: Paroxetine — Anti-depressant
  Arms: Intervention
Drug: Sertraline — Anti-depressant
  Arms: Intervention
Drug: Citalopram — Anti-depressant
  Arms: Intervention
Drug: Venlafaxine — Anti-depressant
  Arms: Intervention
Drug: Duloxetine — Anti-depressant
  Arms: Intervention
Drug: Mirtazapine — Anti-depressant
  Arms: Intervention
Drug: Diphenhydramine — Sleep medication
  Arms: Intervention
Drug: Trazodone — Sleep medication
  Arms: Intervention
Drug: Prazosin — Sleep medication
  Arms: Intervention

SUMMARY:
The overarching goal of this UH2-UH3 proposal is to work with the NIH Health Care Systems Research Collaboratory to develop and implement a large scale, cluster randomized pragmatic clinical trial demonstration project that directly informs national trauma care system policy targeting injured patients with presentations of Posttraumatic Stress Disorder (PTSD) and related comorbidity. Each year in the United States (US), over 30 million individuals present to trauma centers, emergency departments, and other acute care medical settings for the treatment of physical injuries. Multiple chronic conditions including enduring PTSD, alcohol and drug use problems, depression and associated suicidal ideation, pain and somatic symptom amplification, and chronic medical conditions (e.g., hypertension, coronary artery disease, diabetes, and pulmonary diseases) are endemic among physical trauma survivors with and without traumatic brain injuries (TBI). Evidence-based, collaborative care/care management treatment models for PTSD and related comorbidities exist. These care management models have the potential to be flexibly implemented in order to prevent the development of chronic PTSD and depressive symptoms, alcohol use problems, and enduring physical disability in survivors of both TBI and non-TBI injuries; care management models may also be effective in mitigating the impact of the acute injury event on symptom exacerbations in the large subpopulation of injury survivors who already carry a substantial pre-injury burden of multiple chronic medical conditions.

DETAILED DESCRIPTION:
Primary Aims and Hypotheses

The primary aim of the UH3 period is to conduct a pragmatic randomized effectiveness trial of a collaborative care intervention targeting PTSD and comorbid conditions after acute care injury hospitalization. The investigation aims to determine if injured patients receiving the collaborative care intervention demonstrate significant reductions in PTSD symptoms when compared to control patients receiving care as usual. The study also aims to determine if the intervention patients when compared to control patients will demonstrate significant reductions in depressive symptoms, suicidal ideation, and alcohol use problems, and improvements in physical function. The primary hypothesis is that the intervention group when compared to the control group will demonstrate significant reductions in PTSD symptoms over the course of the year after injury. Secondary hypotheses are that intervention patients when compared to control patients will demonstrate, significant reductions in depressive symptoms, significant reductions in alcohol use problems, and improved post-injury physical function.

A Priori Secondary Analyses

The study team hypothesizes that a subgroup of patients will have persistent PTSD symptoms that will not remit over the longitudinal course of the investigation, regardless of randomization to intervention or control group conditions. The study team also anticipates that readily identifiable baseline clinical, injury and demographic characteristics will be associated with persistent PTSD symptoms over time (e.g., higher PTSD symptom levels, greater pre-injury trauma exposure, intentional injury including firearm related injury mechanisms and other characteristics such as unemployment, as well as other baseline factors). Derived from previous randomized clinical trials, a cumulative burden index has been developed from these baseline characteristics and will be adapted for the current investigation. The study team proposes a series of secondary analyses that adjust for and stratify by baseline characteristics that put patients at risk for persistent symptoms. It is hypothesized that these secondary analyses will identify a subgroup of intervention patients who are not at risk for persistent symptoms and who will demonstrate clinically and statistically significant treatment responses when compared to patients with similar baseline characteristics in the control condition. The study team also hypothesizes that the treatment effects will be greatest at the 1-6 month post-injury time points that are temporally correlated with the period of active intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient currently admitted to inpatient/emergency department for a traumatic injury

Exclusion Criteria:

* Non-English speaking
* Self-inflicted injury
* Actively psychotic
* Incarcerated or in custody
* Less than 35 on PTSD Checklist
* Less than 3 items on PTSD medical record screen
* Less than 2 pieces of contact information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 635 (Actual)
Dates: Start 2015-10; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Zatzick, MD, Principal Investigator — University of Washington
Locations (24):
- United States (24):
  - Honor Health, Scottsdale, Arizona
  - Cedars Sinai, Beverly Hills, California
  - U.C. Davis, Sacramento, California
  - Santa Clara Valley Medical Center, San Jose, California
  - U.C.L.A. Harbor, Torrance, California
  - Hartford Hospital, Hartford, Connecticut
  - Georgia Regents, Augusta, Georgia
  - Eskenazi Health, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Louisiana State University, New Orleans, Louisiana
  - Regions Hospital, Saint Paul, Minnesota
  - University of Rochester, Rochester, New York
  - Jacobi Medical Center, The Bronx, New York
  - Wake Forest, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Baylor Health Care System, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - The University of Utah, Salt Lake City, Utah
  - The University of Vermont, Burlington, Vermont
  - Inova Trauma Center, Falls Church, Virginia
  - The University of Wisconsin Madison, Madison, Wisconsin

REFERENCES:
- [Derived] Abu K, Bedard-Gilligan M, Moodliar R, Bulger EM, Hernandez A, Knutzen T, Shoyer J, Birk N, Conde C, Engstrom A, Ryan P, Wang J, Russo J, Zatzick DF. Can stepped collaborative care interventions improve post-traumatic stress disorder symptoms for racial and ethnic minority injury survivors? Trauma Surg Acute Care Open. 2024 Jan 24;9(1):e001232. doi: 10.1136/tsaco-2023-001232. eCollection 2024. PMID 38287923
- [Derived] Zatzick D, Palinkas L, Chambers DA, Whiteside L, Moloney K, Engstrom A, Prater L, Russo J, Wang J, Abu K, Iles-Shih M, Bulger E. Integrating pragmatic and implementation science randomized clinical trial approaches: a PRagmatic Explanatory Continuum Indicator Summary-2 (PRECIS-2) analysis. Trials. 2023 Apr 21;24(1):288. doi: 10.1186/s13063-023-07313-0. PMID 37085877
- [Derived] Nguyen J, Whiteside LK, Bulger EM, Veach L, Moloney K, Russo J, Nehra D, Wang J, Zatzick DF. Post-traumatic stress disorder (PTSD) symptoms and alcohol and drug use comorbidity at 25 US level I trauma centers. Trauma Surg Acute Care Open. 2022 Aug 4;7(1):e000913. doi: 10.1136/tsaco-2022-000913. eCollection 2022. PMID 35979039
- [Derived] Engstrom A, Moloney K, Nguyen J, Parker L, Roberts M, Moodliar R, Russo J, Wang J, Scheuer H, Zatzick D. A Pragmatic Clinical Trial Approach to Assessing and Monitoring Suicidal Ideation: Results from A National US Trauma Care System Study. Psychiatry. 2022 Spring;85(1):13-29. doi: 10.1080/00332747.2021.1991200. Epub 2021 Dec 21. PMID 34932440
- [Derived] Nehra D, Bulger EM, Maier RV, Moloney KE, Russo J, Wang J, Anderson K, Zatzick DF. A Prospective US National Trauma Center Study of Firearm Injury Survivors Weapon Carriage and Posttraumatic Stress Disorder Symptoms. Ann Surg. 2021 Oct 1;274(4):e364-e369. doi: 10.1097/SLA.0000000000005043. PMID 34225296
- [Derived] Zatzick D, Jurkovich G, Heagerty P, Russo J, Darnell D, Parker L, Roberts MK, Moodliar R, Engstrom A, Wang J, Bulger E, Whiteside L, Nehra D, Palinkas LA, Moloney K, Maier R. Stepped Collaborative Care Targeting Posttraumatic Stress Disorder Symptoms and Comorbidity for US Trauma Care Systems: A Randomized Clinical Trial. JAMA Surg. 2021 May 1;156(5):430-474. doi: 10.1001/jamasurg.2021.0131. PMID 33688908
- [Derived] Zatzick DF, Russo J, Darnell D, Chambers DA, Palinkas L, Van Eaton E, Wang J, Ingraham LM, Guiney R, Heagerty P, Comstock B, Whiteside LK, Jurkovich G. An effectiveness-implementation hybrid trial study protocol targeting posttraumatic stress disorder and comorbidity. Implement Sci. 2016 Apr 30;11:58. doi: 10.1186/s13012-016-0424-4. PMID 27130272

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: The intervention aims to prevent the development of chronic PTSD and depressive symptoms, alcohol use problems, and enduring physical disability in survivors of both traumatic brain injury(TBI) and non-TBI injuries. The intervention utilizes a computerized decision support tool to flexibly target these multiple conditions including and includes care management, motivational interviewing, cognitive behavioral therapy elements, psychotropic drugs, and psychotherapy elements.
  Motivational Interviewing
  Cognitive Behavioral Therapy Elements
  Care Management
  Fluoxetine: Anti-depressant
  Fluvoxamine: Anti-depressant
  Paroxetine: Anti-depressant
  Sertraline: Anti-depressant
  Citalopram: Anti-depressant
  Venlafaxine: Anti-depressant
  Duloxetine: Anti-depressant
  Mirtazapine: Anti-depressant
  Diphenhydramine: Sleep medication
  Trazodone: Sleep medication
  Prazosin: Sleep medication
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 265 | 370
Completed | 188 | 289
Not Completed | 77 | 81

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 265 | 370 | 635
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (13.4) | 39.9 (14.8) | 39.0 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 161 | 308
  Male | 118 | 209 | 327
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 52 | 102
  Not Hispanic or Latino | 214 | 316 | 530
  Unknown or Not Reported | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 127 | 188 | 315
  Race: Black | 89 | 129 | 218
  Race: American Indian | 6 | 9 | 15
  Race: Asian | 2 | 2 | 4
  Race: Pacific Islander | 3 | 1 | 4
  Race: Mixed | 11 | 9 | 20
  Race: Other | 27 | 32 | 59
Baseline PCL-C total score [Mean (Standard Deviation); unit: units on a scale] — The investigators will use the PTSD Checklist - Civilian (PCL-C). The scoring of the scale ranges from a minimum of 17 to a maximum of 85, with higher scores indicating a worse outcome. The measure can also provide a rating of symptoms consistent with a diagnosis of PTSD.
  units on a scale | 54.0 (12.6) | 50.7 (11.2) | 52.1 (11.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline PTSD Checklist- Civilian (PCL-C) Over the Course of the Year After Injury
Description: The investigators will use the PTSD Checklist - Civilian (PCL-C). The scoring of the scale ranges from a minimum of 17 to a maximum of 85, with higher scores indicating a worse outcome. The measure can also provide a rating of symptoms consistent with a diagnosis of PTSD.
Time Frame: Baseline, 3-month, 6-month, 12-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 265 | 370
score on a scale
  Change from Baseline at 3 Months | -1.65 (0.86) | 0.08 (0.74)
  Change from Baseline at 6 Months | -4.02 (0.99) | -1.44 (0.83)
  Change from Baseline at 12 Months | -5.51 (1.18) | -4.25 (0.97)

2. Primary Outcome: Change From Baseline Patient Health Questionnaire 9 Item Depression Scale Over the Course of the Year After Injury
Description: The investigators will use the Patient Health Questionnaire 9-item Depression Scale (PHQ-9). The scoring of the scale ranges from a minimum of 0 to a maximum of 27, with higher scores indicating a worse outcome.
Time Frame: Baseline, 3-month, 6-month, 12-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 265 | 370
score on a scale
  Change from Baseline at 3 Months | -0.79 (0.40) | -0.50 (0.35)
  Change from Baseline at 6 Months | -1.17 (0.45) | -0.90 (0.38)
  Change from Baseline at 12 Months | -1.84 (0.52) | -2.16 (0.43)

3. Primary Outcome: Change From Baseline Alcohol Use Disorders Identification Over the Course of the Year After Injury
Description: The investigators will use the Alcohol Use Disorders Identification Test (AUDIT) as a continuous measure. The 10-item scale score ranges from 0-40, with higher values indicating a worse outcome.
Time Frame: Baseline, 3-month, 6-month, 12-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 265 | 370
score on a scale
  Change from Baseline at 3 Months | -2.04 (0.21) | -1.90 (0.18)
  Change from Baseline at 6 Months | -1.69 (0.22) | -1.63 (0.19)
  Change from Baseline at 12 Months | -1.81 (0.23) | -1.45 (0.19)

4. Primary Outcome: Change From Baseline Short Form (SF)-12/36 Physical Function Over the Course of the Year After Injury
Description: The investigators used the Medical Outcomes Study Short Form healthy survey (MOS SF-12/36) physical components summary to assess physical function. The minimum and maximum scores are 0-100 with higher scores representing a better outcome.
Time Frame: Baseline, 3-month, 6-month, 12-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 265 | 370
score on a scale
  Change from Baseline at 3 Months | -16.78 (0.69) | -15.90 (0.59)
  Change from Baseline at 6 Months | -14.17 (0.79) | -13.83 (0.66)
  Change from Baseline at 12 Months | -13.23 (0.94) | -11.68 (0.77)

5. Secondary Outcome: Number of Participants With Suicidal Ideation
Description: Item 9 of the Patient Health Questionnaire 9-item (PHQ-9) scale assesses suicidal ideation. It is scored from 0 to 3, with a score of 1 or greater indicating a patient has suicidal ideation. Participants with a PHQ-9 item 9 score of greater than or equal to 1 are reported for this outcome.
Time Frame: Baseline, 3-month, 6-month, 12-month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 265 | 370
Participants
  Baseline | 67 | 90
  3 Month | 69 | 99
  6 Month | 63 | 106
  12 Month | 51 | 92

6. Secondary Outcome: Number of Participants Endorsing a Single Item That Assesses Opioid Use
Description: Single items that assess non-prescribed opioid use. Single item self-report dichotomized as none versus at least monthly use.
Time Frame: Baseline, 3-month, 6-month, 12-month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 265 | 370
Participants
  Baseline | 18 | 44
  3 Month | 4 | 15
  6 Month | 4 | 20
  12 Month | 6 | 6

7. Secondary Outcome: Cognitive Impairment Scale
Description: The investigators will use the National Study on the Costs and Outcomes of Trauma (NSCOT) Cognitive Screen, a 4 - Item Traumatic Brain Injury / Post-concussive Symptom Screen. The scoring of the scale ranges from a minimum of 4 to a maximum of 20, with lower scores indicating a worse outcome.
Time Frame: Baseline, 3-month, 6-month, 12-month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 265 | 370
score on a scale
  Baseline | 13.5 (4.6) | 13.4 (4.5)
  3 Month | 13.3 (4.5) | 13.2 (4.5)
  6 Month | 13.2 (4.7) | 13.4 (4.1)
  12 Month | 13.8 (4.7) | 14.2 (4.1)

8. Secondary Outcome: Brief Pain Inventory
Description: A brief measure scored on a 0 to 10 scale to assess a patient's pain, with a higher score indicating more severe pain; a score of 0 indicates no pain and a score of 10 indicates very severe pain.
Time Frame: Baseline, 3-month, 6-month, 12-month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 265 | 370
score on a scale
  Baseline | 6.8 (2.4) | 6.7 (2.7)
  3 Month | 4.3 (2.9) | 4.7 (2.8)
  6 Month | 4.1 (3.1) | 4.5 (3.0)
  12 Month | 3.9 (3.0) | 3.8 (3.0)

9. Secondary Outcome: SF-36 Quality of Life
Description: The SF-36 assess quality of life domains that span emotional health, overall health status, and role function; a score of 100 indicates perfect health and a score of 0 indicates extremely poor health.
Time Frame: Baseline, 3-month, 6-month, 12-month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 265 | 370
score on a scale
  Baseline | 44.3 (13.9) | 45.1 (13.0)
  3 Month | 38.3 (12.4) | 39.1 (13.0)
  6 Month | 38.4 (14.0) | 39.5 (12.2)
  12 Month | 39.2 (13.6) | 41.4 (11.9)

10. Secondary Outcome: TSOS Patient Satisfaction: Overall Health Care
Description: Satisfaction with health care was rated on a scale of 1 to 5, with 1 indicating very dissatisfied and 5 indicating very satisfied.
Time Frame: Baseline, 3-month, 6-month, 12-month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 265 | 370
score on a scale
  Baseline | 4.4 (0.9) | 4.4 (0.9)
  3 Month | 3.9 (1.1) | 3.8 (1.1)
  6 Month | 4.0 (1.1) | 3.8 (1.1)
  12 Month | 3.9 (1.1) | 3.8 (1.2)

11. Secondary Outcome: Number of Participants Endorsing a Single Item That Assesses Stimulant Use
Description: Single items that assess non-prescribed stimulant use. Single item self-report dichotomized as none versus at least monthly use.
Time Frame: Baseline, 3-month, 6-month, 12-month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 265 | 370
Participants
  Baseline | 58 | 77
  3 Month | 9 | 17
  6 Month | 7 | 22
  12 Month | 8 | 16

12. Secondary Outcome: Number of Participants Endorsing a Single Item That Assesses Marijuana Use
Description: Single items that assess marijuana use. Single item self-report dichotomized as none versus at least monthly use.
Time Frame: Baseline, 3-month, 6-month, 12-month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 265 | 370
Participants
  Baseline | 125 | 177
  3 Month | 60 | 72
  6 Month | 60 | 82
  12 Month | 51 | 79

13. Secondary Outcome: TSOS Patient Satisfaction: Mental Health Care
Description: Satisfaction with mental health care was rated on a scale of 1 to 5, with 1 indicating very dissatisfied and 5 indicating very satisfied.
Time Frame: Baseline, 3 Month, 6 Month, 12 Month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 265 | 370
score on a scale
  Baseline | 4.1 (1.0) | 4.0 (1.1)
  3 Month | 3.6 (1.1) | 3.5 (1.1)
  6 Month | 3.6 (1.1) | 3.4 (4.1)
  12 Month | 3.7 (1.1) | 3.5 (1.1)

ADVERSE EVENTS:
Time Frame: Baseline, 3 Month, 6 Month, and 12 Month
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 6/265 | 3/370
Serious Adverse Events (participants affected / at risk) | 15/265 | 13/370
Other Adverse Events (participants affected / at risk) | 134/265 | 197/370
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=265) | Usual Care (N=370)
Suicide Attempt (Injury, poisoning and procedural complications) | 9 | 10
Death (General disorders) | 6 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=265) | Usual Care (N=370)
Suicidal Ideation (Psychiatric disorders) | 134 | 197

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT02655354/Prot_SAP_000.pdf